CLINICAL TRIAL: NCT03914404
Title: A 12-week, Multi-center, Randomized, Double-blind, Double Dummy, Parallel Clinical Trial to Compare the Efficacy of γ-linolenic Acid and Thioctic Acid in Patients With Diabetic Neuropathy
Brief Title: Efficacy of γ-linolenic Acid and Thioctic Acid in Patients With Diabetic Neuropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Tae Sun Park, Obesity Research Center of Chonbuk National University, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DLB-DN-EVOP
Record Dates: First submitted 2019-04-10; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Diabetic Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Thioctic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): * γ-linoleic acid (Evoprim soft capsule) twice a day and 4 capsules at a time.
  * Thioctic Acid(LipoA HR Tab. 600mg) placebo once a day and 1 tablet at a time.
  Interventions: Drug: γ-linoleic acid and placebo(Thioctic Acid)
- Control Group (Experimental): * Thioctic Acid(LipoA HR Tab. 600mg) once a day and 1 tablet at a time.
  * γ-linoleic acid (Evoprim soft capsule) placebo twice a day and 4 capsules at a time.
  Interventions: Drug: Thioctic Acid and placebo(γ-linoleic acid)

INTERVENTIONS:
Drug: γ-linoleic acid and placebo(Thioctic Acid) — * γ-linoleic acid (Evoprim soft capsule) twice a day and 4 capsules at a time.
  * Thioctic Acid(LipoA HR Tab. 600mg) placebo once a day and 1 tablet at a time.
  Arms: Test group
Drug: Thioctic Acid and placebo(γ-linoleic acid) — * Thioctic Acid(LipoA HR Tab. 600mg) once a day and 1 tablet at a time.
  * γ-linoleic acid (Evoprim soft capsule) placebo twice a day and 4 capsules at a time.
  Arms: Control Group

SUMMARY:
This study was a 12-week, multi-center, randomized, double-blind, double dummy, parallel clinical trial to compare the efficacy of γ-linolenic acid and Thioctic acid in patients with diabetic neuropathy.

DETAILED DESCRIPTION:
This study evaluated non-inferiority about the efficacy and safety of γ-linolenic acid (Evoprim soft capsule) through patients with diabetic neuropathy were compared γ-linolenic acid (Evoprim soft capsule) and Thioctic acid(LipoA HR Tab. 600mg) using double-blind, double dummy clinical trials. First outcome measures are Visual Analog Scale(VAS) and Total Symptom Score(TSS), secondary outcome measures are Michigan Neuropathy Screening Instrument(MNSI), Current perception Threshold(CPT), Modified Brief Pain Inventory-diabetic polyneuropathy(Modified BPI-DPN) and EuroQol-5 Dimensions(EQ 5D).

ELIGIBILITY:
Inclusion Criteria:

* Patients who were between 20 years and 75 years at screening
* Patients who were diagnosed with type 2 diabetes and whose HbA1c levels were less than 11% at screening
* Patients with a score of 4 or more on the Visual Analogue Score(VAS)
* One or more of the following items

  * If the physical examination score of the Michigan Neuropathy Screening Instrument Score (MNSI) is more than 2 points at the initial screening
  * type 2 diabetic patient who complained one or more of pain, burning sensation, numbness, and sensory loss and measured the current perception threshold (CPT) of the peroneal nerve at three frequencies (2000Hz, 250Hz, 5Hz) Anyone whose diabetes mellitus has been diagnosed as diabetic neuropathy
* Patients who decided to voluntarily participate in clinical trials and agreed in writing

Exclusion Criteria:

* Peripheral neuropathy caused by other causes other than diabetes
* Those are suffering from other painful conditions that are so severe that diabetic neuropathy can not be assessed
* If you have a progressive or degenerative neurological disorder
* Patients with a systolic blood pressure(SBP)≥ 160 mmHg or ≤ 100 mmHg or a diastolic blood pressure(DBP) ≥ 95 mmHg or ≤ 60 mmHg
* Patients who were positive for human immunodeficiency virus (HIV), hepatitis B (HBV), or hepatitis C (HCV) test
* patients with liver dysfunction (ALT / AST> 3 times the upper limit of normal)
* Patients with renal dysfunction (Serum creatine> 2.0 mg / dl)
* Patients with thyroid dysfunction (Thyroid and anti-thyroid medications may be included in this study if they are maintained in normal state.)
* Patients with amputation (including toes) or infections of the lower extremities
* The following diseases are clinically significant patients

  * Unstable coronary artery disease or peripheral vascular disease
  * Liver, kidney, lung, hematologic disease
  * Cancer (within 5 years if possible)
* Patients who have suicide attempts or suicidal tendencies and who have a psychiatric history within 6 months before starting the trial
* Patients with substance abuse or chronic alcohol abuse within 2 years prior to taking the test
* Patients who received intravenous steroid injection or topical anesthetic injection within 2 months before participating in the study
* Patients who participated in other studies within 4 weeks before participating in the trial, or who are currently taking medication for other research
* Screening After randomization for 2 weeks (pause period) before screening, antipsychotics, antipsychotics, sleep depressants, antidepressants, antiepileptics, muscle relaxants, analgesics (narcotic analgesics, NSAIDs, tramadol etc.) Patients who received capsaicin or who received percutaneous electrical nerve stimulation therapy (TENS) or acupuncture
* Patients with a history of hypersensitivity or clinically significant hypersensitivity reactions to this drug substance and soybean oil, soy or peanut
* Patients with clinically significant skin disease or severe skin irritability
* Pregnant or lactating women
* patients suffering from schizophrenia or those who are treated with chloropromazine, mesoridazine, thioridazine, fluphenazine, perphenazine, trifluoperazine, haloperidol (haloperidol), loxapine (loxapine) and other drugs known to cause epileptic seizures
* In addition to the above items, patients who are deemed inappropriate by clinical trial researchers

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-01-26 (Actual); Primary Completion 2016-03-30 (Actual); Study Completion 2018-07-25 (Actual)

PRIMARY OUTCOMES:
Changes of Visual Analog Scale(VAS) | 12 weeks
  The Visual Analog Scale(VAS) score is 0 point for no symptom, 10 points for the most severe symptom, and the patient is asked to mark the degree of subjective pain symptoms as an integer.
Changes of Total Symptom Score(TSS) | 12 weeks
  Total Symptom Score(TSS) classifies diabetic neuropathy symptoms into four categories (pain, burning pain, paresthesia, numbness). The frequency (Occasional, Frequent, Continuous) and symptom intensity (Absent, Slight, Moderate, Severe) are calculated through each question and the score is obtained according to the visual analog scale. It is calculated from 0 point up to 14.64 points.

SECONDARY OUTCOMES:
Changes of Michigan Neuropathy Screening Instrument(MNSIQ) | 12 weeks
  A 15-item questionnaire (MNSIQ) is used to assess deformation, infection, skin thickening of the skin's stratum corneum, and ulcers.
  MNSIQ was designed to screen for diabetic neuropathy through questionnaires on 15 questions that are related to neuropathic symptoms (pain, temperature, and sensation). Two of 15 (number 4 and 10) are vascular symptoms and are excluded from the total score regardless of the results. If you answered 'No' to questions 7 and 13, you will get 1 point. In the end, scores ranging from 0 to 13 indicate that the higher the score, the more severe the neuropathic symptoms.
Changes of Michigan Neuropathy Screening Instrument(MNSIE) | 12 weeks
  A foot test (MNSIE) is used to assess deformation, infection, skin thickening of the skin's stratum corneum, and ulcers.
  MNSIE evaluates foot shape, foot ulceration, ankle reflex, sense of vibration of big toe, monofilament right and left. The score ranges from point 0 to 10, and when the score is above 2, it is diagnosed as neuropathy.
Changes of Current perception Threshold(CPT) | 12 weeks
  Sensory nerve conduction threshold (SNCT) is a unique method for evaluating all three sensory neurons (small unmyelinated fibers, small myelinated fibers, and large myelinated fibers) that make up more than 90% of sensory nerves. It seems to be possible to objectively evaluate sensory nerve of small fiber which recovered early in diabetic neuropathy(Using neurometer).
Changes of Modified Brief Pain Inventory-diabetic polyneuropathy(Modified BPI-DPN) | 12 weeks
  Modified Brief Pain Inventory-diabetic polyneuropathy(Modified BPI-DPN) displays the pain area on the human figure, the number of pain sites, treatment of pain, and pain medication.
  Pain severity refers to the pain sensation- identification aspect (pain threshold). The worst pain, the least pain, the pain average, and the pain now for the last 24 hours are displayed on the 10-point scale (0 points: none, ~ 10 Point: too big to imagine). Pain interference is the emotional-synchronous aspect of pain (pain tolerance). It classifies general activity, mood, walking, working, relationship, sleep and enjoyment of life, and use the 10-point scale (0 points: none to 10 points: completely disturbed).
Changes of EuroQol-5 Dimensions(EQ 5D) | 12 weeks
  EQ-5D index = 1 - (0.050 + 0.096 M2 + 0.418 x M3 + 0.046 x SC2 + 0.13 x SC3 + 0.051 x UA2 + 0.028 x UA3 + 0.037 x PD2 + 0.151 x PD3 + 0.043 x AD2 + 0.158 x AD3 + 0.050 × N3) - 1 if the variable is applicable, 0 if not (M: mobility, SC: self-care, UA: usual activity,, PD: pain / discomfort, AD: anxiety / depression)
  * Variable definition
  * M2: 1 if mobility is 'level 2', 0 if not
  * M3: 1 if mobility is 'level 3', 0 if not
  * SC2: 1 if self-care is 'level 2', 0 if not
  * SC3: 1 if self-care is 'level 3', 0 if not
  * UA2: 1 if usual activity is 'level 2', 0 if not
  * UA3: 1 if usual activity is 'level 3', 0 if not
  * PD2: 1 if pain / discomfort is 'level 2', 0 if not
  * PD3: 1 if pain / discomfort is 'level 3', 0 if not
  * AD2: 1 if anxiety / depression is 'level 2', 0 if not
  * AD3: 1 if anxiety / depression is 'level 3', 0 if not
  * N3: 1 if there is at least one level 3, others are 0

CONTACTS AND LOCATIONS:
Overall Officials: Bong-Yeon Cha, MD,PhD, Principal Investigator — The Catholic University of Korea; Jong hwa Kim, MD, Principal Investigator — Sejong General Hospital; Lee-byeong Park, MD,PhD, Principal Investigator — Gachon University Gil Medical Center; Hyuk Sang Kwon, MD,PhD, Principal Investigator — The catholic university of korea Yeouido st. mary's hospital; In Joo Kim, MD,PhD, Principal Investigator — Pusan National University Hospital; Ji hyun Lee, MD,PhD, Principal Investigator — Daegu Catholic University Medical Center; sung soo Moon, MD,PhD, Principal Investigator — DongGuk University; Sung wan Chun, MD,PhD, Principal Investigator — Soon Chun Hyang University; Byung-Wan Lee, MD,PhD, Principal Investigator — Yonsei univesity severance hospital; Jong chul Won, MD,PhD, Principal Investigator — Inje University; Tae-Sun Park, MD,PhD, Principal Investigator — Chonbuk National University Hospital
Locations (11):
- South Korea (11):
  - Sejong hospital, Bucheon-si, Gyeonggi-do
  - Obesity Research Center of Chonbuk National University, Jeonju, Jeollabuk-do
  - Dongguk university gyeongju hospital, Gyeongju, North Gyeongsang-do
  - Soon chun hyang university hospital cheonan, Cheonan, South Chungcheong Province
  - Daegu Catholic University Medical Center, Daegu
  - Gachon University Gil Medical Center, Incheon
  - Pusan National University Hospital, Pusan
  - Inje university sanggye paik hospital, Seoul
  - Yonsei univesity severance hospital, Seoul
  - The catholic university of korea seoul st. mary's hospital, Seoul
  - The catholic university of korea Yeouido st. mary's hospital, Seoul